CLINICAL TRIAL: NCT06255652
Title: Oral Versus Intravenous Antibiotic Prophylaxis Before Obstetric and Gynecological Procedures
Status: Recruiting | Type: Observational
Sponsor: Sohag University (Other)
Collaborators: Randers Regional Hospital (Other)
Responsible Party: Principal Investigator, Yasmin Tharwat Anwar, Resident of obstetric and gynecology department, Sohag University Hospitals, Sohag University
Other Study IDs: Soh-Med-23-09-05MS
Record Dates: First submitted 2024-02-05; First posted 2024-02-13 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Site Infection
Keywords: SSI
MeSH Terms: interventions — Cephradine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Obstetrician and gynaecological procedures: Patients for obstetricians
  Interventions: Drug: Cephradin

INTERVENTIONS:
Drug: Cephradin — Velosef
  Other Names: Velosef

SUMMARY:
Oral versus intravenous antimicrobial prophylaxis for the prevention of surgical site infection for elective cesarean section and gynacological procedures

DETAILED DESCRIPTION:
the aim of the current study is to compare the efficacy of prophylactic intravenous (cephradine) and oral antibiotic (cephradine) for the prevention of surgical site infection in the elective obctetric and gynecological procedures

ELIGIBILITY:
Inclusion Criteria:

- Cesarean section Gynaecological procedure Exclusion Criteria Immunocompromised patient

-

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: Female patient Pregnant For gynaecological procedure
Sampling Method: Non-Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
proportion of patients with any SSI within 30 days after surgery | July 2024
  July 2024

CONTACTS AND LOCATIONS:
Overall Officials: Hatem Awaga Awaga, Doctor, Study Director — Sohag University
Locations (1):
- Sohag university hospital, Sohag, Egypt

REFERENCES:
- [Derived] Elftooh Awaga HA, Anwar YT, Ait-Allah AS, Abdelkareem AO. Oral versus intravenous antibiotic prophylaxis before obstetric and gynecological surgical interventions: A randomized clinical trial. Eur J Obstet Gynecol Reprod Biol. 2025 Jul;311:114020. doi: 10.1016/j.ejogrb.2025.114020. Epub 2025 Apr 29. PMID 40334373